CLINICAL TRIAL: NCT04226703
Title: The Role of Indirect Laryngoscopy, Clinical and Ultrasonographic Assessment in Prediction of Difficult Airway
Brief Title: Indirect Laryngoscopy and Ultrasonography in Prediction of Difficult Airway
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Hakan Kara, Resident, Istanbul University
Other Study IDs: 2019/722
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Difficult Intubation
Keywords: airway; laryngoscopy; ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients over the age of 18 who underwent surgery in the ear, nose and throat department.
  Interventions: Diagnostic Test: Ultrasonographic upper airway measurements

INTERVENTIONS:
Diagnostic Test: Ultrasonographic upper airway measurements — Ultrasonographic upper airway measurements: Epiglottis-skin distance, Hyoid bone-skin distance, Anterior commissure-skin distance and Thickness of tounge root.
  Indirect Laryngoscopy: Grading of laryngoscopic view (I=Visible anterior commissure and vocal cords, II= visible posterior part of vocal cords and posterior commissure, III= Visible posterior commissure and epiglottis, IV= Visible only epiglottis tip and posterior pharyngeal wall)
  Other Names: Indirect Laryngoscopy

SUMMARY:
This study was designed to assess the success of indirect laryngoscopy and ultrasonographic measurements in the prediction of difficult airway. All patients were examined by indirect laryngoscopy and ultrasonography preoperatively and the predictive values for difficult airway of these methods were compared.

DETAILED DESCRIPTION:
Difficult airway is a condition that increases the patient's vital risk and leaves the anesthesia and surgical team in a difficult position. Failure to perform an adequate preoperative evaluation may result in the team being unprepared. Therefore, various methods have been investigated in the prediction of difficult airway from past to present. With the development of technology, imaging methods have become routine applications in clinical use. Ultrasonography and indirect laryngoscopy have been shown to be used in predicting difficult airway in the literature, but there is no study showing which is a better predictor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is operated in ear, nose and throat department.
* Subject over the age of 18.
* Subject giving consent to participate in the study.

Exclusion Criteria:

* Subject under the age of 18
* Subject with a history of radiotherapy in the head and neck region,
* Subject with facial deformity,
* Subject whose neck movements have been restricted by previous trauma or surgery,
* Subject has laryngeal disease
* Previously operated subject with known airway assessment
* Morbidly obese subject with BMI> 40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who apply to ear, nose and throat department for any kind of otorhinolaryngological operation are included into the study.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Cormack-Lehane Classification | Three minutes after induction of anesthesia.
  The anesthesiologist, who is blind about indirect laryngoscopy findings and ultrasonographic airway measurements, performs intubation and evaluates the laryngeal view.
Epiglottis skin distance in centimeters. | Five minutes before induction of anesthesia.
  The anesthesiologist, who is blind about indirect laryngoscopy findings and is experienced user of ultrasonography, measures epiglottis to skin distance.
Hyoid bone-skin distance in centimeters. | Five minutes before induction of anesthesia.
  The anesthesiologist, who is blind about indirect laryngoscopy findings and is experienced user of ultrasonography, measures hyoid bone to skin distance.
Anterior commissure-skin distance in centimeters. | Five minutes before induction of anesthesia.
  The anesthesiologist, who is blind about indirect laryngoscopy findings and is experienced user of ultrasonography, measures anterior commissure to skin distance.
Thickness of tongue root in centimeters. | Five minutes before induction of anesthesia.
  The anesthesiologist, who is blind about indirect laryngoscopy findings and is experienced user of ultrasonography, measures thickness of tongue root.
Indirect Laryngoscopic Grade | The day before surgery
  The otolaryngologist,who is blind about ultrasonographic airway measurements of patients, performs indirect laryngoscopy and evaluates the laryngeal view.

SECONDARY OUTCOMES:
Body mass index (BMI) | The day before surgery
  Weight and height will be combined to report BMI in kg/m^2.Evaluated by the anesthesiologist who performs intubation.
Thyromental distance in centimeters | The day before surgery
  The distance between thyroid notch and mentum. Evaluated by the anesthesiologist who performs intubation.
Sternomental distance in centimeters. | The day before surgery
  The distance between sternal notch and mentum. Evaluated by the anesthesiologist who performs intubation.
Neck circumference in centimeters. | The day before surgery
  Evaluated by the anesthesiologist who performs intubation.
Mallampati classification | The day before surgery
  Evaluated by the anesthesiologist who performs intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Başaran, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parameswari A, Govind M, Vakamudi M. Correlation between preoperative ultrasonographic airway assessment and laryngoscopic view in adult patients: A prospective study. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):353-358. doi: 10.4103/joacp.JOACP_166_17. PMID 29109635
- [Background] Sanchez-Morillo J, Estruch-Perez MJ, Hernandez-Cadiz MJ, Tamarit-Conejeros JM, Gomez-Diago L, Richart-Aznar M. Indirect laryngoscopy with rigid 70-degree laryngoscope as a predictor of difficult direct laryngoscopy. Acta Otorrinolaringol Esp. 2012 Jul-Aug;63(4):272-9. doi: 10.1016/j.otorri.2012.01.007. Epub 2012 Mar 17. English, Spanish. PMID 22425162